CLINICAL TRIAL: NCT06312020
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of HZN-1116 in Participants With Sjögren's Syndrome
Brief Title: A Phase 2 Study to Investigate Efficacy and Safety of HZN-1116 in Participants With Sjogren's Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-HZN-1116-201
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Sjogren's Syndrome
Keywords: SS; Sjogren's; HZN-1116; Autoimmune disease; Dry Eye syndrome; VIB1116
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- HZN-1116 Dose 1 in Population 1 (Experimental): Participants will receive Dose 1 of HZN-1116
  Interventions: Drug: HZN-1116
- HZN-1116 Dose 2 in Population 1 (Experimental): Participants will receive Dose 2 of HZN-1116
  Interventions: Drug: HZN-1116
- Placebo in Population 1 (Placebo Comparator): Participants will receive Placebo matched to HZN-1116
  Interventions: Drug: Placebo
- HZN-1116 Dose 1 in Population 2 (Experimental): Participants will receive Dose 1 of HZN-1116
  Interventions: Drug: HZN-1116
- HZN-1116 Dose 2 in Population 2 (Experimental): Participants will receive Dose 2 of HZN-1116
  Interventions: Drug: HZN-1116
- HZN-1116 Dose 3 in Population 2 (Experimental): Participants will receive Dose 3 of HZN-1116
  Interventions: Drug: HZN-1116
- HZN-1116 Dose 4 in Population 2 (Experimental): Participants will receive Dose 4 of HZN-1116
  Interventions: Drug: HZN-1116
- Placebo in Population 2 (Placebo Comparator): Participants will receive Placebo matched to HZN-1116
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HZN-1116 — Subcutaneous Administration
  Other Names: VIB1116; AMG 329; Adezkibart
  Arms: HZN-1116 Dose 1 in Population 1; HZN-1116 Dose 1 in Population 2; HZN-1116 Dose 2 in Population 1; HZN-1116 Dose 2 in Population 2; HZN-1116 Dose 3 in Population 2; HZN-1116 Dose 4 in Population 2
Drug: Placebo — Subcutaneous Administration
  Arms: Placebo in Population 1; Placebo in Population 2

SUMMARY:
The purpose of this study is to measure the efficacy and safety of HZN-1116 in participants with Sjogren's syndrome (SS).

DETAILED DESCRIPTION:
The study will enroll 2 SS populations: Population 1 will include participants with moderate to high systemic disease activity; Population 2 will include participants with moderate to severe subjective symptoms. This study will include 3 periods: screening (5 weeks), treatment period (48 Weeks) and follow-up period (12 weeks). In the treatment period, participants from each of the populations will be randomized to receive subcutaneous (SC) dose of HZN-1116 or placebo.

Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with SS by meeting the 2016 American College of Rheumatology (ACR)/EULAR Classification Criteria.
* Have an ESSDAI score of >= 5 at screening (only for Population 1).
* Have an ESSPRI score of >= 5 at screening (only for Population 2).
* Have an ESSDAI score of < 5 at screening (only for Population 2).
* Positive for anti-Ro autoantibodies, rheumatoid factor (RF) at screening, or both at screening.

Key Exclusion Criteria:

* Concomitant system sclerosis.
* Active malignancy or history of malignancy within the last 5 years with exception of in situ carcinoma of the cervix treated with apparent success with curative therapy > 12 months prior to screening; OR cutaneous basal cell carcinoma following presumed curative therapy.
* Individuals who are pregnant or lactating or planning to become pregnant during the study.
* Individuals who have a positive test for, or have been treated for, hepatitis B, hepatitis C, or HIV infection.
* Individuals with history of more than one episode of herpes zoster and/or opportunistic infections in the last 12 months, with the exception of non-invasive herpes simplex at any site, oral candidiasis, vaginal candidiasis, or cutaneous fungal infections, which are permitted within the prior 12 months unless of unusual severity. Individuals with a prior history of ophthalmic herpes zoster will be excluded.
* Active infections requiring systemic treatment at the time of screening or through randomization, or history of more than 2 infections requiring intravenous (IV) antibiotics within 12 months prior to screening.
* Last administration of experimental biologic or oral agents < 6 months or 5 half-lives, whichever is longer, before screening.
* Individuals who have had previous treatment with any biologic B cell-depleting therapy (eg, rituximab, ocrelizumab, inebilizumab, or ofatumumab) within 12 months or other B cell targeting therapy (eg, belimumab) or anti-type I IFN pathway therapy (eg, anifrolumab) < 6 months before randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in European Alliance of Associations for Rheumatology (EULAR) Sjogren's Syndrome Disease Activity Index (ESSDAI) (Population #1) | At Week 48
Change from baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) (Population #2) | At Week 24

SECONDARY OUTCOMES:
Change from baseline in ESSDAI (Population #1) | At Week 24
Proportion of Participants achieving ESSDAI [5] response (Population #1) | At Week 24 and Week 48
Change from baseline in ESSPRI pain domain score (Population #1) | At Week 24 and Week 48
Change from baseline in Diary for Assessing Sjogren's Patient-Reported Outcome Index (DASPRI) pain domain score (Population #1) | At Week 24 and Week 48
Change from baseline in ESSPRI fatigue domain score (Population #1) | At Week 24 and Week 48
Change from baseline in DASPRI fatigue domain score (Population #1) | At Week 24 and Week 48
Change from baseline in ESSPRI dryness domain score (Population #1) | At Week 24 and Week 48
Change from baseline in DASSPRI dryness domain score (Population #1) | At Week 24 and Week 48
Change from baseline in tender joint count (TJC) (Population #1) | At Week 24 and Week 48
Change from baseline in swollen joint count (SJC) (Population #1) | At Week 24 and Week 48
Change from baseline in 36-item Short Form Survey (SF-36) physical component score (PCS) (Population #1) | At Week 24 and Week 48
Change from baseline in 36-item Short Form Survey (SF-36) mental component score (MCS) (Population #1) | At Week 24 and Week 48
Change from baseline in patient-reported outcomes measurement information system (PROMIS)-Fatigue SF-10a (Population #1) | At Week 24 and Week 48
Change from baseline in DASPRI (Population #2) | At Week 24
Proportion of Participants achieving ESSPRI [1.5] response (Population #2) | At Week 24
Change from baseline in ESSPRI pain domain (Population #2) | At Week 24
Change from baseline in ESSPRI fatigue domain (Population #2) | At Week 24
Change from baseline in ESSPRI dryness domain (Population #2) | At Week 24
Change from baseline in SF-36 PCS Score (Population #2) | At Week 24
Change from baseline in 36-item Short Form Survey (SF-36) mental component score MCS (Population #2) | At Week 24
Change from baseline in PROMIS-Fatigue SF-10a (Population #2) | At Week 24
Serum concentration of HZN-1116 starting at Week 1 through study completion (Population #1 and #2) | Up to Week 60
Proportion of Participants who develop anti drug antibodies (ADA) over time (Population #1 and #2) | Up to Week 60

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (65):
- United States (16):
  - Arizona Arthritis & Rheumatology Research-S Vineyard Ave, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Associates -4550 E Bell Rd, Phoenix, Arizona
  - Neurovations Research, Napa, California
  - Life Arc Research Centers Corp, Miami, Florida
  - IRIS Research and Development LLC, Plantation, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Augusta University Medical Center-Augusta-1120 15th St, Augusta, Georgia
  - Tufts Medical Center - 800 Washington St - PPDS, Boston, Massachusetts
  - Pioneer Clinical Research NY, New York, New York
  - DJL Clinical Research PLLC-431 N Wendover Rd, Charlotte, North Carolina
  - Altoona Center for Clinical Research - 175 Meadowbrook Ln, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Tekton Research, LLC - W Gate Blvd - Austin - PPDS, Austin, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - R & H Clinical Research-777 S Fry Rd, Katy, Texas
  - University Of Wisconsin - Madison, Madison, Wisconsin
- Argentina (5):
  - MR Medicina Reumatologica, San Fernando, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Privado de Medicina Familiar, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Buenos Aires, Ciudad Autónoma de BuenosAires
- LKH-Universitätsklinikum Graz - Auenbruggerplatz 15, Graz, Styria, Austria
- Chile (4):
  - Centro de especialidades médicas Vanguardia, Temuco, Región de la Araucanía
  - Centro de Investigacion de Enfermedades Respiratorias e inmunologicas, Viña del Mar, Región de Valparaíso
  - Biomedica Research Group, Providencia, Región-MetropolitanadeSantiago
  - Prosalud y Cia Ltda., Santiago, Región-MetropolitanadeSantiago
- Colombia (4):
  - Centro Integral de Reumatologia del Caribe S.A.S - CIRCARIBE S.A.S., Barranquilla, Atlántico
  - Healthy Medical Center S.A.S., Zipaquirá, Cundinamarca
  - Servimed S.A.S, Bucaramanga
  - AES - AS - Fundacion Centro de Investigacion Clinica - CIC, Medellín
- CHU de Montpellier - Hôpital Lapeyronie, Montpellier, Hérault, France
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Mvz Rheumatologie Und Autoimmunmedizin Hamburg Gmbh, Hamburg
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen, Hajdú-Bihar
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet - Albert Flórián út 5-7, Budapest
- Italy (2):
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome, Lazio
  - IRCCS Ospedale Galeazzi - Sant'Ambrogio, Milan, Lombardy
- Mexico (2):
  - PanAmerican Clinical Research - Domingo Sarmiento 2784 - PPDS, Guadalajara, Jalisco
  - Clinstile, S.A. de C.V., Mexico City
- Poland (10):
  - Pratia Poznan - PPDS, Poznan, Greater Poland Voivodeship
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne PROMED, Krakow, Lesser Poland Voivodeship
  - MICS Centrum Medyczne Warszawa - MICS - PPDS, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. El. Reicher- Spartanska 1, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - FutureMeds - Targowek - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. Z o.o., Malbork, Pomeranian Voivodeship
  - FutureMeds - Krakow - PPDS, Krakow
- Portugal (3):
  - ULS de Santa Maria,EPE - Hospital de Santa Maria - PPDS, Lisbon
  - Hospital Conde de Bertiandos - Unidade Local de saúde do Alto Minho, EPE - Ponte de Lima, Ponte de Lima
  - ULS de Santo António, EPE - Hospital de Santo António, Porto
- Spain (6):
  - Hospital Sanitas CIMA, Barcelona
  - Hospital General Universitario de Castellon, Castellon
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Clinicas Gaias-Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quironsalud Sagrado Corazon, Seville
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- Taiwan (5):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital - PPDS, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com